# Pain sensitization in patients with symptomatic atrial fibrillation compared with asymptomatic patients

Anna Björkenheim, MD, PhD<sup>1</sup>, Adam Jackson, BSc<sup>1</sup> Ole Fröbert, MD, PhD<sup>1</sup>, Dennis Boye Larsen BSc PhD<sup>2</sup>, Lars Arendt Nielsen, MSci, PhD, DMSci<sup>2</sup>

- 1. Department of Cardiology, Faculty of Medicine and Health, Örebro University, Sweden.
- 2. SMI, Faculty of Medicine, Aalborg University, Aalborg, Denmark.

#### **Correspondence:**

Anna Björkenheim, MD, PhD Ole Fröbert, MD, PhD

Department of Cardiology Department of Cardiology

Örebro University Hospital Örebro University Hospital

701 85 Örebro, Sweden 701 85 Örebro, Sweden

Telephone +46 19 602 54 59 Telephone +46 602 54 13

Fax +46 19 602 24 07 Fax +46 19 602 54 38

Date: 2020-11-24

**Abstract** 

Background

Atrial fibrillation (AF) is the most common sustained arrhythmia and the number of patients

with AF is expected to increase substantially in the coming decades. One third of patients

with AF report no AF-associated symptoms, but up to one fourth report severe symptoms

such as chest pain. It is well recognized, but unclear why patients' experience of AF-related

symptoms, including chest pain, varies so much. Patients with chronic pain show a high

degree of central sensitization, i.e. facilitated pain responses to repeated painful stimulation

and impaired conditioned pain modulation, compared with controls. It is possible that

patients with symptomatic AF may have developed pronounced pain sensitization even in

the absence of chest pain as a symptom. No previous study has investigated pain

sensitization in patients with AF.

**Objective and methods** 

The primary objective is to assess differences in pain sensitization in patients with

symptomatic AF compared with patients with asymptomatic AF. Secondary objectives are to

study the association of age, sex, AF duration, comorbidities and health-related quality of life

to pain sensitization. A total of 30 patients with permanent AF (15 symptomatic and 15

asymptomatic) will be recruited. Patients will complete an AF-specific symptom score and a

generic health-related quality of life questionnaire, and physicians will assess AF-related

symptoms. Quantitative sensory testing recordings will be collected by pressure algometry.

Assessment of temporal summation of pressure pain and conditioning pain modulation will

be used to investigate the involvement of pain sensitization.

Clinical relevance

Date:

2020-11-24

Version: 1.2

This preliminary pilot study will be used to estimate sample size for a larger study in which

both patients and control subjects will be recruited, to further investigate whether patients

with symptomatic AF have increased pain sensitization compared with patients with

asymptomatic AF and controls. The studies may have an impact on individualized

management of patients with AF in the future.

**Trial registration** 

The study protocol is registered with ClinicalTrials.gov (NCT...)

Keywords

Atrial fibrillation, Symptoms, Quality of life, Pain, Conditioning pain modulation, Temporal

summation

Date: 2020-11-24


# **Abbreviations**

AF Atrial fibrillation

AF6 Atrial fibrillation 6 questionnaire

CPM Conditioned pain modulation

ECG Electrocardiogram

SF-36 Short form 36 health survey

VAS Visual analogue scale

Date: 2020-11-24

## Introduction

### Background

Atrial fibrillation (AF) is the most common sustained arrhythmia affecting approximately 3% of adults aged 20 years or older in Western countries, and is expected to increase further in the coming decades(1). The presence of AF is independently associated with an increased risk of all-cause mortality and morbidity, largely due to stroke and heart failure, dementia, symptoms, and impaired quality of life(2-7). The management of AF aims to prevent AF-related complications using oral anticoagulation therapy in patients with a high risk of stroke and to reduce symptoms and improve health-related quality of life using a rate (slowing of the ventricular rate) or rhythm control (restoration and maintenance of normal sinus rhythm) strategy(8).

About one third of patients with AF report no AF-associated symptoms, but up to one fourth of patients report severe symptoms such as palpitations, dyspnea, chest discomfort or pain, dizziness and syncope(9-11). In previous studies 9 to 15% of patients with permanent AF reported chest pain as an AF-related symptom(12, 13). In addition, one third of patients with symptomatic AF suffer from psychological distress (anxiety and/or depression), which may also worsen symptoms of AF(11, 14).

It is well recognized, but remains unclear why some patients with AF are asymptomatic whereas others are severely symptomatic. Several studies have evaluated the relationship between patient characteristics and the presence of AF symptoms, and have found that asymptomatic AF is more frequent in men than in women, and in older age(15, 16). Inconsistent results have been reported for associations between asymptomatic AF and comorbidities(17). Patients with all types of AF can be asymptomatic, but asymptomatic AF

Date: 2020-11-24

is more common in patients with permanent AF(18). The situation is further complicated by

the fact that asymptomatic AF episodes are common even in highly symptomatic patients

and that AF interventions such as pulmonary vein isolation increase asymptomatic

episodes(19). In conclusion, little is known of the pathophysiological mechanisms underlying

AF symptomatology but both somatic and psychological factors are likely involved.

The authors have previously shown that central nervous system responses to visceral and

somatosensory nociceptive input are altered in patients who have angina despite normal

coronary angiograms compared to healthy volunteers (20). Patients with chronic pain

conditions such as osteoarthrosis, chronic pancreatitis and irritable bowel syndrome, show a

high degree of central sensitization, i.e. facilitated pain responses to repeated painful

stimulation and impaired conditioned pain modulation (CPM) compared with controls(21-

24). Furthermore, these patients often show a discrepancy between pain intensity and

objective measures of disease severity and healthcare personnel often underestimate

patients' pain intensity(25, 26). It is also well-known that stress influences pain sensitivity

and has been correlated to hyperalgesia in patients with ischemic heart disease(27, 28). It is

possible that patients with symptomatic AF have developed pronounced pain sensitization

even in the absence of chest pain as a symptom, and in particular facilitated pain responses

to repeated painful stimulation, i.e. temporal summation of pressure pain. No previous

study has investigated pain sensitization in patients with AF, neither in patients with or

without chest pain as a symptom.

**Purpose** 

Date:

2020-11-24


The primary objective is to assess differences in pain sensitization in patients with

symptomatic AF compared with patients with asymptomatic AF.

**Hypothesis** 

We hypothesize that central sensitization is involved in sensing of and discomfort from AF in

symptomatic patients, involving neural pathways also involved in perceiving pain. Because of

shared pathways, we further hypothesize that patients with AF symptoms have lower pain

thresholds than asymptomatic patients with AF.

**Clinical relevance** 

It is well recognized, but unclear why patients' perception of AF varies so much. This

preliminary pilot trial will be used to estimate sample size for a larger trial, in which both

patients and control subjects will be recruited, to further investigate whether patients with

symptomatic AF have increased pain sensitization compared with patients with

asymptomatic AF and controls. The studies may have an impact on individualized

management of patients with AF in the future.

Date: 2020-11-24


**Material and methods** 

Study design

Single-center cohort study.

Subject inclusion criteria

Study participants will be recruited from a database of all patients aged 20 years or older

with a diagnosis of AF from 1 January 2015 to 31 December 2018 in Örebro County (more

than 10 000 patients) extracted from the National Patient Register, that covers all in-patient

and outpatient physician visits from both private and public caregivers, and the Medrave 4

patient statistics software that is used in all public general practices in the county. The

diagnosis of AF was based on at least one electrocardiogram (ECG) characterized by an

absolutely irregular RR interval, no distinct P waves and an atrial cycle length of less than 200

ms. By accepted convention, an episode with these ECG characteristics lasting for at least 30

seconds was diagnostic of AF(8). Permanent AF is defined as persistent AF that is accepted

by both the patient and the physician and for which no further attempts to restore or

maintain normal sinus rhythm will be undertaken(8).

Further inclusion criteria:

- Male or female subjects  $\geq$  20 years and  $\leq$  75 year, primarily 60 to 70 years old.

- Permanent AF

- Previously completed AF-specific symptoms questionnaire Atrial fibrillation 6

questionnaire (AF6)

- Written informed consent

Subject exclusion criteria

Date:

2020-11-24

Date.


- Paroxysmal or persistent AF (AF that terminates spontaneously or with intervention,

respectively(8))

Previous pulmonary vein isolation

Psychiatric or cognitive condition

Pregnancy

Previous/current drug or alcohol abuse

- Previous neurological or concomitant musculoskeletal disorders

- Continuous analgesic medication

**Examinations** 

All potential patients will receive written information about the study and will thereafter be

contacted by telephone and offered an outpatient visit to a physician at the Department of

cardiology, Örebro University Hospital, Örebro, Sweden. After obtaining written informed

consent, patients will be asked to complete the AF6 and the Short form 36 health survey (SF-

36) questionnaires before a 12-lead ECG is obtained. Patients will also be asked to rate the

symptom chest pain on the Visual analogue scale (VAS) (0 to 10) and to draw the pain area

on a body chart. Comorbidities, medications and duration of AF will be documented and a

routine clinical examination will be performed, and the modified European Heart Rhythm

Association symptoms scale assessed. Quantitative sensory testing recordings will be

collected by pressure algometry. The patients will be asked not to take any analgesic

medication 24 hours before the examination. No follow-up visits are scheduled. Subjects will

be divided into two groups based on their previous AF6 symptom scores; asymptomatic

patients with an AF6 sum score of 0, and symptomatic patients with an AF6 sum score of

≥30.

Date:

2020-11-24


Symptom assessment

The patient-reported AF6 questionnaire includes six items (breathing difficulties at rest and

upon exertion, limitations in day-to-day life, feeling of discomfort, tiredness and

worry/anxiety due to AF) and a score of 0 (no symptoms) to 10 (severe symptoms) is

reported for each item, and all scores are added into a single sum score. Sum scores range

from 0 to 60, with higher values reflecting more severe AF-related symptoms. The AF6

includes a recall period of the last 7 days(29, 30).

The physician-assessed modified European Heart Rhythm Association symptoms scale is

used for symptom severity assessment in patients with AF, relating specifically to the time

when patients feel symptoms of AF. Patients in class I are considered to have no symptoms,

in class IIa mild, class IIb moderate, class III severe and in class IV disabling symptoms of

AF(8, 31).

Health-related quality of life

The patient-reported SF-36 has a recall period of four weeks and consists of 36 items

assessing eight domains ranging from 0 to 100, with higher values indicating better health-

related quality of life. The eight domains generate two summary measures: the physical

component summary and the mental component summary scores, which will be used to

assess health-related quality of life(32).

**Clinical examination** 

Date:

2020-11-24


A cardiovascular examination including blood pressure measurement will be performed. The

blood pressure will be measured after 15 minutes of rest by an automatic

sphygmomanometer.

Quantitative sensory testing

Pressure pain threshold

The pressure pain thresholds (PPTs) is defined as the minimal amount of pressure where a

sense of pressure first changes to pain. Participants will be instructed to press the 'stop'

button of the algometer as soon as the pressure results in the first sensation of pain.

Pressure will be increased at a rate of approximately 30 kPa/s. The 1-cm<sup>2</sup> probe of the

handheld pressure algometer (Somedic AB, Sweden) will be placed perpendicularly to the

skin. PPTs will be assessed over the sternum at the level of intercostal spaces 3-5 and over

the tibia bone(27). The PPTs will be measured three times on each site, and the mean of the

three measurements will be used for statistical analysis. Low PPTs indicate sensitization.

Temporal summation of pressure pain

A Pin prick (tip area, 0.2mm<sup>2</sup>) with a weighted load (Aalborg University, Denmark) will be

used to induce temporal summation of pressure pain (TSP) as previously conducted in other

pain studies(33-35). A force of 50 g will be applied once over the sternum at the level of

intercostal spaces 3–5 and over the tibia bone and the patient will be asked to rate the pain

intensity on the VAS (0 to 10). Then 10 consecutive stimuli will be applied (1 s interval

between consecutive stimuli) to the same site and the subject will be asked to rate the pain

intensity of the last stimulation on the VAS. TSP will be calculated as the difference in the

Date:

2020-11-24


pain intensity between the first and the last stimulation. High TSP scores indicate facilitated

temporal summation.

**Conditioning pain modulation** 

The right hand up to the wrist will be immersed into stirred cold water (2–4 °C, measured in

the water) for 2 min (the so called cold pressor test). Before the immersion the PPTs will be

assessed from the sternum and the tibial bone, at the end of the two min immersion the

PPTs will be assessed again and this will be repeated again 10 min after the hand is

withdrawn from the water. The conditioning pain modulation index will be assessed as the

increase in PPTs during the immersion as compared to the pre-immersion PPTs. The lower

the difference is the more sensitization.

**Primary endpoint** 

The primary objective is to assess differences in pain sensitization in patients with

symptomatic AF compared with patients with asymptomatic AF.

**Secondary endpoint** 

Secondary objectives are to study the association of age, sex, AF duration and comorbidities

and physical and mental component summary scores to pain sensitization.

**Ethics approval** 

The study protocol is approved by the Swedish Ethical Review Authority (2020-01619).

Statistics and data management

Date:

2020-11-24


Data collected during the study will be coded.

Statistical analysis

Data will be presented as mean and standard deviation. A one-way ANOVA will be used for

demographic parameters and to compare the groups. Pearson correlations will be used for

linear estimates and Spearman's correlations for non-linear parameters. All analyses will be

adjusted for age. Analyses will be performed using IBM SPSS Statistics 22 (Armonk, NY, USA)

or STATA release 14 (College Station, TX, USA).

Sample size calculations

As no previous trial of pain sensitization in patients with AF has been performed, a pilot trial

is necessary to calculate sample size for a larger study.

**Database and Case report form** 

A case report form will be filled out and coded for each patient. The investigators are

responsible for ensuring the accuracy, completeness, legibility and timeliness of the data

recorded in the case report forms.

Documentation and data collection

Criteria for inclusion, informed consent, the decision to include the subject and the subject

number will be documented in the subject's hospital record.

Insurance

The subjects in the study are covered by the Swedish patient insurances.

**Economy** 

The trial is an academic study conceived and conducted by healthcare personnel. The study

is independent of commercial interests. Study logistics, handling of data and statistical

Date:

2020-11-24


assessment will be financed by the Department of Cardiology, Örebro University Hospital,

Sweden. The investigators will apply for grants from public funds.

**Ethical considerations** 

The study will be conducted in accordance with the Declaration of Helsinki. The cold pressor

test activates the sympathetic nervous system and increases blood pressure and heart rate,

and there is a slight risk of angina during the test. There are otherwise no known risks or

complications associated with the quantitative sensory testing but it may cause some

temporary mild to moderate discomfort.

The patient is free to stop the testing at any time, and in case of angina the testing will be

stopped and the patient will be closely monitored and administered sublingual nitroglycerin.

Risks, side effects, advantages and disadvantages in participation

Subjects will be treated according to standard clinical practice. There is a slight risk of the

test causing angina chest pain. However, we do not expect that subjects will have any

disadvantages from participating in the study. The risk of complications during quantitative

sensory testing is considered low.

Guidelines for obtaining informed consent

Subjects will enter the study after signing the informed consent form. Candidate participants

will receive written information of the study, and oral information by a physician

participating in the study. The subjects will be given time to think through participation in

the study and to ask questions. Informed consent will be obtained by a Good Clinical Practice

qualified physician participating in the study.

Withdrawal

Date:

2020-11-24


A subject can withdraw from the study at any time. Data collected up to the end of follow-up

will be used in the final analysis of the study.

**Publication** 

Results, positive as well as negative or inconclusive, will be published in an international

medical journal, primarily in a cardiology journal.

End of trial and archiving

The study will end when the last subject has signed informed consent, completed the

questionnaires and has undergone clinical examination and quantitative sensory testing. The

steering committee reserves the right to terminate the study prematurely e.g. if the study

participant recruitment is too slow, if study participant retention in the study is insufficient

or if undue risk related to the quantitative sensory testing arises. Data collected during the

study will be archived for at least 10 years after the study has been completed.

Date: 2020-11-24


#### References

- 1. Zoni-Berisso M, Lercari F, Carazza T, Domenicucci S. Epidemiology of atrial fibrillation: European perspective. (1179-1349 (Print)).
- 2. Bjorck S, Palaszewski B Fau Friberg L, Friberg L Fau Bergfeldt L, Bergfeldt L. Atrial fibrillation, stroke risk, and warfarin therapy revisited: a population-based study. (1524-4628 (Electronic)).
- 3. Haim M, Hoshen M, Reges O, Rabi Y, Balicer R, Leibowitz M. Prospective national study of the prevalence, incidence, management and outcome of a large contemporary cohort of patients with incident non-valvular atrial fibrillation. (2047-9980 (Electronic)).
- 4. Benjamin EJ, Wolf Pa Fau D'Agostino RB, D'Agostino Rb Fau Silbershatz H, Silbershatz H Fau Kannel WB, Kannel Wb Fau Levy D, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. (0009-7322 (Print)).
- 5. Stewart S, Hart Cl Fau Hole DJ, Hole Dj Fau McMurray JJV, McMurray JJ. A population-based study of the long-term risks associated with atrial fibrillation: 20-year follow-up of the Renfrew/Paisley study. (0002-9343 (Print)).
- 6. Thrall G, Lane D Fau Carroll D, Carroll D Fau Lip GYH, Lip GY. Quality of life in patients with atrial fibrillation: a systematic review. (1555-7162 (Electronic)).
- 7. Jacobs V, Cutler MJ, Day JD, Bunch TJ. Atrial fibrillation and dementia. (1873-2615 (Electronic)).
- 8. Kirchhof P Fau Benussi S, Benussi S Fau Kotecha D, Kotecha D Fau Ahlsson A, Ahlsson A Fau Atar D, Atar D Fau Casadei B, Casadei B Fau Castella M, et al. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. (1522-9645 (Electronic)).
- 9. Savelieva I, Camm AJ. Clinical relevance of silent atrial fibrillation: prevalence, prognosis, quality of life, and management. (1383-875X (Print)).
- 10. Patel N, Chung EH, Mounsey JP, Schwartz JD, Pursell I, Gehi AK. Effectiveness of atrial fibrillation monitor characteristics to predict severity of symptoms of atrial fibrillation. (1879-1913 (Electronic)).
- 11. Thrall G, Lip Gy Fau Carroll D, Carroll D Fau Lane D, Lane D. Depression, anxiety, and quality of life in patients with atrial fibrillation. (0012-3692 (Print)).
- 12. Lip GY, Laroche C, Ioachim PM, Rasmussen LH, Vitali-Serdoz L, Petrescu L, et al. Prognosis and treatment of atrial fibrillation patients by European cardiologists: one year follow-up of the EURObservational Research Programme-Atrial Fibrillation General Registry Pilot Phase (EORP-AF Pilot registry). (1522-9645 (Electronic)).
- 13. Nabauer M, Gerth A Fau Limbourg T, Limbourg T Fau Schneider S, Schneider S Fau Oeff M, Oeff M Fau Kirchhof P, Kirchhof P Fau Goette A, et al. The Registry of the German Competence NETwork on Atrial Fibrillation: patient characteristics and initial management. (1532-2092 (Electronic)).
- 14. Lane DA, Langman Cm Fau Lip GYH, Lip Gy Fau Nouwen A, Nouwen A. Illness perceptions, affective response, and health-related quality of life in patients with atrial fibrillation. (0022-3999 (Print)).
- 15. Walfridsson UA-Ohoo, Steen Hansen P, Charitakis EA-Ohoo, Almroth H, Jonsson A, Karlsson LOA-Ohoo, et al. Gender and age differences in symptoms and health-related quality of life in patients with atrial fibrillation referred for catheter ablation. (1540-8159 (Electronic)).
- 16. Reynolds MR, Lavelle T Fau Essebag V, Essebag V Fau Cohen DJ, Cohen DJ Fau Zimetbaum P, Zimetbaum P. Influence of age, sex, and atrial fibrillation recurrence on quality of life outcomes in a population of patients with new-onset atrial fibrillation: the Fibrillation Registry Assessing Costs, Therapies, Adverse events and Lifestyle (FRACTAL) study. (1097-6744 (Electronic)).

Date: 2020-11-24

- 17. Ballatore A, Matta M, Saglietto A, Desalvo P, Bocchino PP, Gaita F, et al. Subclinical and Asymptomatic Atrial Fibrillation: Current Evidence and Unsolved Questions in Clinical Practice. LID E497 [pii] LID 10.3390/medicina55080497 [doi]. (1648-9144 (Electronic)).
- 18. Rienstra M, Lubitz Sa Fau Mahida S, Mahida S Fau Magnani JW, Magnani JW Fau Fontes JD, Fontes Jd Fau Sinner MF, Sinner Mf Fau Van Gelder IC, et al. Symptoms and functional status of patients with atrial fibrillation: state of the art and future research opportunities. (1524-4539 (Electronic)).
- 19. Hindricks G, Piorkowski C Fau Tanner H, Tanner H Fau Kobza R, Kobza R Fau Gerds-Li J-H, Gerds-Li Jh Fau Carbucicchio C, Carbucicchio C Fau Kottkamp H, et al. Perception of atrial fibrillation before and after radiofrequency catheter ablation: relevance of asymptomatic arrhythmia recurrence. (1524-4539 (Electronic)).
- 20. Frobert O, Arendt-Nielsen L Fau Bak P, Bak P Fau Funch-Jensen P, Funch-Jensen P Fau Peder Bagger J, Peder Bagger J. Pain perception and brain evoked potentials in patients with angina despite normal coronary angiograms. (1355-6037 (Print)).
- 21. Arendt-Nielsen L, Nie H Fau Laursen MB, Laursen Mb Fau Laursen BS, Laursen Bs Fau Madeleine P, Madeleine P Fau Simonsen OH, Simonsen Oh Fau Graven-Nielsen T, et al. Sensitization in patients with painful knee osteoarthritis. (1872-6623 (Electronic)).
- 22. Staud R, Cannon Rc Fau Mauderli AP, Mauderli Ap Fau Robinson ME, Robinson Me Fau Price DD, Price Dd Fau Vierck CJ, Jr., Vierck CJ, Jr. Temporal summation of pain from mechanical stimulation of muscle tissue in normal controls and subjects with fibromyalgia syndrome. (0304-3959 (Print)).
- 23. Sandrini G, Rossi P Fau Milanov I, Milanov I Fau Serrao M, Serrao M Fau Cecchini AP, Cecchini Ap Fau Nappi G, Nappi G. Abnormal modulatory influence of diffuse noxious inhibitory controls in migraine and chronic tension-type headache patients. (0333-1024 (Print)).
- 24. Olesen SS, Brock C Fau Krarup AL, Krarup Al Fau Funch-Jensen P, Funch-Jensen P Fau Arendt-Nielsen L, Arendt-Nielsen L Fau Wilder-Smith OH, Wilder-Smith Oh Fau Drewes AM, et al. Descending inhibitory pain modulation is impaired in patients with chronic pancreatitis. (1542-7714 (Electronic)).
- 25. Arendt-Nielsen L, Morlion B, Perrot S, Dahan A, Dickenson A, Kress HG, et al. Assessment and manifestation of central sensitisation across different chronic pain conditions. (1532-2149 (Electronic)).
- 26. Puntillo K, Neighbor M Fau O'Neil N, O'Neil N Fau Nixon R, Nixon R. Accuracy of emergency nurses in assessment of patients' pain. (1524-9042 (Print)).
- 27. Bergmann N, Ballegaard S Fau Holmager P, Holmager P Fau Kristiansen J, Kristiansen J Fau Gyntelberg F, Gyntelberg F Fau Andersen LJ, Andersen LJ Fau Hjalmarson A, et al. Pressure pain sensitivity: a new method of stress measurement in patients with ischemic heart disease. (1502-7686 (Electronic)).
- 28. Richebe P Fau Rivat C, Rivat C Fau Cahana A, Cahana A. Stress-induced hyperalgesia: any clinical relevance for the anesthesiologist? (1528-1175 (Electronic)).
- 29. Harden M, Nystrom B Fau Kulich K, Kulich K Fau Carlsson J, Carlsson J Fau Bengtson A, Bengtson A Fau Edvardsson N, Edvardsson N. Validity and reliability of a new, short symptom rating scale in patients with persistent atrial fibrillation. (1477-7525 (Electronic)).
- 30. Harden M, Nystrom B Fau Bengtson A, Bengtson A Fau Medin J, Medin J Fau Frison L, Frison L Fau Edvardsson N, Edvardsson N. Responsiveness of AF6, a new, short, validated, atrial fibrillation-specific questionnaire--symptomatic benefit of direct current cardioversion. (1572-8595 (Electronic)).
- 31. Wynn GJ, Todd DM, Webber M, Bonnett L, McShane J, Kirchhof P, et al. The European Heart Rhythm Association symptom classification for atrial fibrillation: validation and improvement through a simple modification. (1532-2092 (Electronic)).

Date: 2020-11-24

- 32. McHorney CA, Ware Je Jr Fau Lu JF, Lu Jf Fau Sherbourne CD, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. (0025-7079 (Print)).
- 33. Petersen KK, Arendt-Nielsen L Fau Simonsen O, Simonsen O Fau Wilder-Smith O, Wilder-Smith O Fau Laursen MB, Laursen MB. Presurgical assessment of temporal summation of pain predicts the development of chronic postoperative pain 12 months after total knee replacement. (1872-6623 (Electronic)).
- 34. Neogi T, Guermazi A, Roemer F, Nevitt MC, Scholz J, Arendt-Nielsen L, et al. Association of Joint Inflammation With Pain Sensitization in Knee Osteoarthritis: The Multicenter Osteoarthritis Study. (2326-5205 (Electronic)).
- 35. Neogi T, Frey-Law L, Scholz J, Niu J, Arendt-Nielsen L, Woolf C, et al. Sensitivity and sensitisation in relation to pain severity in knee osteoarthritis: trait or state? (1468-2060 (Electronic)).

Date: 2020-11-24